CLINICAL TRIAL: NCT05230524
Title: DIAMOND AF Post-Approval Study
Acronym: DAF PAS
Status: Terminated | Type: Observational
Why Stopped: Sponsor and FDA agreed on early termination.
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: DIAMOND AF PAS
Record Dates: First submitted 2022-01-27; First posted 2022-02-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: DiamondTemp™ Ablation System — Pulmonary vein isolation will be performed with the DiamondTemp™ Ablation System

SUMMARY:
The DIAMOND AF Post Approval study is a prospective, global, multi-center, non-randomized, single-arm observational trial

DETAILED DESCRIPTION:
The DIAMOND AF PAS is a prospective, global, multi-center, non-randomized, single-arm observational trial. This post approval study is a condition of the Pre-Market Approval order (P200028/S002) by the U.S. Food and Drug Administration." The purpose of this clinical study is to describe clinical performance and safety data in a broad patient population treated with the DiamondTemp™ Ablation System. To assess clinical performance and safety of the DiamondTemp™ Ablation System, study objectives will estimate primary efficacy through 36 months, and primary procedural safety at 12 months. Additionally, study objectives will characterize the ablation procedure, change in QoL through 36 months, single procedure success rate, freedom from symptomatic recurrence, and adverse events (AE) through 36 months.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of recurrent symptomatic paroxysmal AF
2. Failure or intolerance of at least one Class I or III antiarrhythmic drug (including sotalol)
3. Patient is ≥ 18 years of age
4. Planned procedure for the treatment of AF using commercially available DiamondTemp™ Ablation System
5. Patient is willing and able to provide written informed consent
6. Patient is willing and able to comply with study requirements

Exclusion Criteria:

1. Prior persistent AF (continuous AF that is sustained >7 days)
2. Patient with life expectancy that makes it unlikely 36 months of follow-up will be completed.
3. Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of this study not pre-approved by Medtronic
4. Patients with contraindications to a Holter monitor
5. Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects ≥ 18 years of age who have a recommendation for an ablation with the DiamondTemp™ Ablation System may be approached regarding enrollment in this study.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Freedom from Atrial Fibrillation (AF) /Atrial Flutter (AFL) /Atrial Tachycardia (AT) | 36 month
  Estimate the 36-month freedom from AF/AFL/AT recurrence following ablation procedure using the DiamondTemp™ Ablation System.
Freedom from Primary Safety Events | 12 months
  Estimate primary safety adverse event rate for ablation using the DiamondTemp™ Ablation System through 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Study Director — Medtronic CAS Chief Medical Officer
Locations (5):
- Florida Electrophysiology LLC, Winter Park, Florida, United States
- France (2):
  - Centre Hospitalier de Pau - Hôpital François Mitterrand, Pau
  - Reunion University Hospital - Saint Pierre, Saint-Pierre
- Italy (2):
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti di Ancona, Ancona
  - Humanitas Mater Domini, Varese